CLINICAL TRIAL: NCT04263467
Title: High Intensity Aerobic Exercise Training and Immune Cell Mobilization in Patients With Lung Cancer (HI AIM)
Acronym: HIAIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Per thor Straten, Professor, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LU2006
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Cancer of Lung
MeSH Terms: conditions — Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive a 6-weeks exercise-based intervention with supervised and group-based exercise training three times a week at the hospital setting. Each training session will consist of intermediate and high intensity interval training. The exercise-based intervention will be combined with standard oncological treatments; checkpoint inhibitors, checkpoint inhibitors combined with chemotherapy or oncological surveillance. Additional monitoring of patient will include physical tests, questionnaires and blood samples.
  Interventions: Other: Exercise intervention
- Control group (Experimental): Participants in the control group will receive standard oncological treatments; immune checkpoint inhibitors, checkpoint inhibitors combined with chemotherapy or oncological surveillance. Additional monitoring of patient will include physical tests, questionnaires and blood samples.
  Interventions: Other: Standard oncological treatments

INTERVENTIONS:
Other: Exercise intervention — The exercise intervention will consist a intermediate to high aerobic exercise training program.
  Arms: Intervention group
Other: Standard oncological treatments — Standard oncological treatments
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate if high-intensive training can mobilize and activate the immune system, and thereby enhance the effect of the conventional treatment of lung cancer patients. An important aspect of this study will investigate if the presence of various proteins and cells in blood and tumor biopsies can verify or predict the effect of the high-intensive training. In this clinical trial, patients with lung cancer will combine their conventional therapy with a six-week exercise program.

DETAILED DESCRIPTION:
Research has shown that exercise training has several beneficial effects in cancer patients and survivors both during and after anti-cancer treatment, including improved physical function, reduction of symptoms, reduction of side effects and improved quality of life (QoL). In addition, a physical active lifestyle is associated with reduced risk of some cancers. Recent data in mouse models have shown that tumor-bearing mice randomized to a voluntary wheel running group showed over 60% reduction in tumor incidence and progression in several tumor models. Moreover, the mouse data clearly showed homing of T and natural killer (NK) cells to tumors in an exercise dependent manner, underscoring that exercise may render patients more prone to respond to therapy. However, most of the underlying biological mechanisms leading to the documented beneficial effects of physical exercise in relation to cancer are yet unknown, but exercise-mediated changes in hormone levels, inflammation and immune cell function are thought to play a key role.

Included participants will be randomized 1:1 to an intervention group and a control group. Participants in the intervention group will receive a six-weeks exercise-based intervention with supervised and group-based exercise training three times a week at the hospital setting. Each training session will consist of intermediate and high intensity interval training. The exercise-based intervention will be combined with standard oncological treatments; checkpoint inhibitors, checkpoint inhibitors combined with chemotherapy or oncological surveillance. Participants in the control group will still receive standard oncological treatments; immune checkpoint inhibitors, checkpoint inhibitors combined with chemotherapy or oncological surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic non-small cell lung cancer
* Measurable disease according to RECIST 1.1
* Age ≥ 18 years
* Treatment with immune checkpoint inhibitors, checkpoint inhibitors combined with chemotherapy or oncological surveillance
* Eastern Cooperative Oncology Group (ECOG) performance status score (PS) ≤2
* Preferably metastasis suitable for biopsy
* Normal marrow function as defined below:

  * White blood cell count (WBC) ≥ 2 x 10⁹/L
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
  * Hemoglobin ≥ 6.0 mmol/l
  * Platelet count ≥ 100 x 10⁹/L
  * In case, a patient's bone marrow values fall slightly below the described values, the treatment responsible doctor will be consulted. The general health and the ability to proceed with the treatment will be considered.
* Ability to speak and read Danish
* Willingness to give informed consent for participation in the study

Exclusion Criteria:

* Any physical condition that hinder the execution of physical exercise, as assessed by the referring oncologist and by a physiotherapist
* Severe dyspnea that hinder the execution of high intensity aerobic exercise training, as assessed by the referring oncologist
* Symptomatic brain metastases
* Dementia, psychotic disorders, or other cognitive diseases or conditions that hinder participation in a clinical exercise-based trial, as assessed by the referring oncologist
* Unstable medical disease or history of serious or concurrent illness; any medical condition that might be aggravated by exercise training or that cannot be controlled, including, but not restricted to congestive heart failure (NYHA class III-IV), unstable angina pectoris, implantable cardioverter defibrillator (ICD), or myocardial infarction within 6 months
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications. Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted
* Use of beta blockers
* Any systemic infections within the last 4 weeks
* Patients who receives chemotherapy as monotherapy
* In patients with documented bone metastases; patients with:

  * A bone metastatic burden or location that poses a risk of injury in the performance of exercise training, as assessed by the referring oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Circulating NK cells | 0 - 36 months
  Flow cytometry will be used to analyse and determine amount of circulating NK cells. The analysis will focus on absolute counts of NK cells, but also surface expression of various surface markers of interest.

SECONDARY OUTCOMES:
Maximal aerobic capacity | 0 - 36 months
  Measure difference in maximal aerobic capacity before and after exercise intervention.
Circulating T cells and B cells. | 0 - 36 months
  Flow cytometry will be used to analyse and determine amount of circulating NK cells. The analysis will focus on absolute counts of NK cells, but also surface expression of various surface markers of interest eg. PD-1.
Circulating serum markers of inflammation | 0 - 36 months
  We aim to establish a panel of serum markers that reflect the effect of exercise training. This will be establish through big panel analysis of inflammatory markers using luminex assays. We will compare serum from blood samples taken before and after exercise training.
Overall survival | 0 - 36 months
  Overall Survival (OS), defined as time from treatment initiation to death, will be described with use of Kaplan Meier curve.
Progression free survival (PFS) | 0 - 36 months
  Defined as the time from the date of randomization until the date of progressive disease (PD). This is determined by investigator assessment of objective radiographic disease assessments per Response Evaluation Criteria In Solid Tumors (RECIST 1.1) and immune RECIST (iRECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Per thor Straten, Professor, Study Director — CCIT
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) sharing plan will be consider at the end of the trial.

REFERENCES:
- [Derived] Holmen Olofsson G, Mikkelsen MK, Ragle AM, Christiansen AB, Olsen AP, Heide-Ottosen L, Horsted CB, Pedersen CMS, Engell-Noerregaard L, Lorentzen T, Persson GF, Vinther A, Nielsen DL, Thor Straten P. High Intensity Aerobic exercise training and Immune cell Mobilization in patients with lung cancer (HI AIM)-a randomized controlled trial. BMC Cancer. 2022 Mar 5;22(1):246. doi: 10.1186/s12885-022-09349-y. PMID 35247994